CLINICAL TRIAL: NCT00874965
Title: Study of the Benefits of Lower Limb Electrostimulation Training on Muscular Parameters and Minute Ventilation During Exercise in Severe and Deconditioned COPD Patients.
Brief Title: Electrostimulation, Skeletal Muscle Function, and Exercise Capacity in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: ESTIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Marthe Bélanger, Professionnel de recherche, Laval University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CER20105
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease (COPD); Electrostimulation; Muscle function; Exercise ventilation; Anabolism/catabolism pathway
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ES (Active Comparator): Electrostimulation
  Interventions: Device: Electrostimulation
- Sham ES (Placebo Comparator): Sham stimulation
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Electrostimulation — 50Hz; 0.4 ms; 30 min; 5 times / week
  Arms: ES
Device: Sham stimulation — 30 min; 5 times / week
  Arms: Sham ES

SUMMARY:
This study was designed to test the following hypothesis:

The benefit of electrostimulation training will be greater than sham stimulation training in term of muscle strength and mass (muscle hypertrophy), exercise tolerance, reduction of ventilation during exercise and quality of life in COPD patients

DETAILED DESCRIPTION:
Background: Because it has little impact on ventilatory requirements and dyspnea, muscle electrostimulation appears as a promising alternative to general physical reconditioning in advanced COPD and its feasibility has been confirmed in this population. However, the physiological mechanisms underlying the proposed benefits of electrostimulation training have not been explored.

Objective: To evaluate in COPD patients the physiological mechanisms of changes in exercise tolerance after electrostimulation training.

Method: We propose to conduct a controlled, randomized and double blind clinical trial comparing the efficacy of muscle electrostimulation training of the lower limbs to sham training in 24 patients with COPD. Patients are included in either 6 weeks of electrostimulation training (active treatment group) or 6 weeks of sham electrostimulation. Before and after training, patients perform endurance shuttle walking test, muscle function testing, muscle biopsy, blood sampling and health-related quality of life questionnaire.

Planning analysis: The main outcome will be change in the strength of the quadriceps over the 6-week electrostimulation program. The other end-points will be mid-thigh and calf muscle cross-sectional area, lower limb muscle endurance, ventilation, dyspnea, leg fatigue, operational lung volumes at iso-time and walking time during an endurance shuttle walk, muscle hypertrophying/atrophying pathways and muscle aerobic capacity. For each group, pre- and post-training comparisons will be made using a repeated measures design. The magnitude of the pre- and post-training changes will also compared between both groups with a two-way ANOVA (group, training effect) with repeated measures on the second factor (training effect). A p value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* COPD
* FEV1 < 60% predicted value and FEV1/ FVC < 70%
* 6-minute walking distance < 400 m

Exclusion Criteria:

* Patients suffering from cardiovascular, neurological, skeletal muscle, or any other condition that could alter their capacity to perform the exercise test
* Patients taking systemic corticosteroids on a daily basis (patients having received systemic steroids for the treatment of up to two exacerbations in the preceding year and those on inhaled steroids will be allowed)
* Patients with room air PaO2 < 60 mm Hg will be excluded.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-12; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Change in the strength of the quadriceps over the 6-week electrostimulation program. | 6 to 8 weeks

SECONDARY OUTCOMES:
Ventilation at iso-time during an endurance shuttle walkMuscle | 6 to 8 weeks
hypertrophying/atrophying pathways | 6 to 8 weeks
Muscle aerobic capacity: fibre-typing, oxydative enzymes, muscle capillarization | 6 to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: François Maltais, MD, Principal Investigator — Laval University
Locations (1):
- Hôpital Laval, Québec, Quebec, Canada

REFERENCES:
- [Derived] Vivodtzev I, Debigare R, Gagnon P, Mainguy V, Saey D, Dube A, Pare ME, Belanger M, Maltais F. Functional and muscular effects of neuromuscular electrical stimulation in patients with severe COPD: a randomized clinical trial. Chest. 2012 Mar;141(3):716-725. doi: 10.1378/chest.11-0839. Epub 2011 Nov 23. PMID 22116795